CLINICAL TRIAL: NCT06837506
Title: Ultrasound Guided Rectus Sheath Block Versus Intrathecal Morphine for Postoperative Analgesia in Patients Undergoing Open Total Abdominal Hysterectomy: A Randomized Trial
Brief Title: Ultrasound Guided Rectus Sheath Block Versus Intrathecal Morphine for Postoperative Analgesia in Patients Undergoing Open Total Abdominal Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed, Lecturer of Anesthesia, Intensive care, and pain management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R03/2024/2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound; Rectus Sheath Block; Intrathecal Morphine; Postoperative Analgesia; Total Abdominal Hysterectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block group (Experimental): Patients will receive rectus sheath block (20 ml bilaterally, bupivacaine 0.25%) after induction of general anesthesia.
  Interventions: Drug: Rectus sheath block
- Intrathecal morphine group (Experimental): Patients will receive 150 µg intrathecal morphine after induction of general anesthesia.
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Rectus sheath block — Patients will receive rectus sheath block (20 ml bilaterally, bupivacaine 0.25%) after induction of general anesthesia.
  Other Names: Bupivacaine 0.25%
  Arms: Rectus sheath block group
Drug: Intrathecal morphine — Patients will receive 150 µg intrathecal morphine after induction of general anesthesia.
  Arms: Intrathecal morphine group

SUMMARY:
This study aims to compare the effectiveness and safety of ultrasound-guided rectus sheath block versus intrathecal morphine for postoperative analgesia in patients undergoing open total abdominal hysterectomy.

DETAILED DESCRIPTION:
Effective postoperative analgesia is crucial for enhancing recovery and patient satisfaction following major surgical procedures, such as total abdominal hysterectomy (TAH).

Rectus sheath block (RSB), an ultrasound-guided regional anesthesia technique, involves the injection of local anesthetic into the rectus sheath, providing analgesia to the anterior abdominal wall. RSB is used to block the sensory nerves of the anterior abdominal wall and thereby contributing to pain relief after lower abdominal surgeries.

Intrathecal morphine (ITM) provides a highly effective method of analgesia by delivering the medication directly into the cerebrospinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old.
* American Society of Anesthesiologists (ASA) physical status (I -II).
* Patients undergoing open total abdominal hysterectomy.

Exclusion Criteria:

* Hepatic, renal, or cardiac disease.
* Any known allergy to local anesthetic.
* Physical or mental conditions which may vague measuring postoperative pain following surgery.
* History of chronic use of analgesic as nonsteroidal anti-inflammatory drugs (NSAIDs) or central nervous system (CNS) depressants as antiepileptic, and bleeding disorders.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing open total abdominal hysterectomy
Enrollment: 80 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Morphine will be administered if the visual analog scale (VAS) score is ≥ 4.

SECONDARY OUTCOMES:
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery till first dose of morphine administrated)
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed after surgery over 24 hour using VAS scale at (post-anesthesia care unit, 2, 4, 6, 12, 18, and 24 h).
Degree of sedation | Intraoperatively
  Sedation will be assessed using Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S): (5 Alert: Responds readily to name spoken in normal tone, 4: Lethargic response to name spoken in normal tone, 3: Responds only after name is called loudly and/or repeatedly, 2: Responds only after mild prodding or shaking ,1: Responds only after painful trapezius squeeze,0: Does not respond to painful trapezius squeeze).
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Time of hospital discharge | 28 days postoperatively
  Time of hospital discharge will be recorded from admission till the discharge from hospital.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as hematoma, nerve damage or neuropathy, bradycardia, hypotension, nausea, vomiting, pruritis, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: The data will be available upon a reasonable request from the corresponding author.
Access Criteria: After the end of study for one year.